CLINICAL TRIAL: NCT05198609
Title: Camrelizumab, Apatinib Plus Hepatic Arterial Infusion Chemotherapy Versus Camrelizumab and Apatinib for Hepatocellular Carcinoma With Portal Vein Invasion: a Randomized, Open-label, Multicentre Trial
Brief Title: Camrelizumab, Apatinib Plus HAIC Versus Camrelizumab and Apatinib for HCC With Portal Vein Invasion: a Randomized Trial
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: First People's Hospital of Foshan (Other); Zhongshan People's Hospital, Guangdong, China (Other); Affiliated Hospital of Guangdong Medical University (Other); Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Shi Ming, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-HCC-II-013
Record Dates: First submitted 2021-12-29; First posted 2022-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma, hepatic arterial infusion chemotherapy, immunotherapy, targeted therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Camrelizumab, Apatinib Plus FOLFOX-HAIC (Experimental)
  Interventions: Procedure: FOLFOX-HAIC; Drug: Camrelizumab; Drug: Apatinib
- Camrelizumab and Apatinib (Active Comparator)
  Interventions: Drug: Camrelizumab; Drug: Apatinib

INTERVENTIONS:
Procedure: FOLFOX-HAIC — Hepatic arterial infusion of oxaliplatin (85mg/m2,IA,day 1, hour 0-2), fluorouracil (400mg/m2,IA,day 1, hour 3), leucovorin (400mg/m2, IV,day 1, hour 2-3) and fluorouracil (2400mg/m2, IA, hour 3-23) repeated every 4 weeks for a total of six times
  Arms: Camrelizumab, Apatinib Plus FOLFOX-HAIC
Drug: Camrelizumab — Camrelizumab was administered 200mg intravenously for 30-60 minutes every 2 weeks, and the maximum cumulative duration of Camrelizumab is 2 years. The shortest time interval between two administrations should not be less than 12 days.
Drug: Apatinib — Apatinib was administered orally 250mg once per day

SUMMARY:
Compare the efficacy and safety of camrelizumab, apatinib plus FOLFOX-HAIC and camrelizumab plus apatinib in hepatocellular carcinoma with portal vein invasion.

ELIGIBILITY:
Inclusion Criteria:

1. volunteered with written inform consent
2. unresectable HCC or progression after surgery or locoregional threapy, with the diagnosis confirmed by histologic or cytologic analysis or clinical features according to the American Association for the Study of Liver Diseases practice guidelines and the China liver cancer (CNLC) guidelines
3. Patients with portal vein tumor thrombosis (PVTT) confirmed by 2 kinds of imaging examinations
4. no previous systemic therapy for HCC. Herbs, Chinese medicines or proprietary Chinese medicines that contain anti-cancer active ingredients in the instructions are allowed, but such treatments need to be terminated before randomization
5. at least 1 measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
6. patients who had previously received local treatments (such as radiofrequency ablation, percutaneous ethanol or acetic acid injection, cryoablation, high-intensity focused ultrasound, trans-arterial chemoembolization, trans-arterial embolization, etc.)were allowed to be enrolled, but it was required that the target lesions were with no previous local treatment, or the target lesion had received local treatment but had progression according to the RECIST v1.1
7. an Eastern Cooperative Oncology Group performance status of 0 to 1
8. Child-Pugh A class liver function
9. adequate organ function (absoluteneutrophil count ≥1.5 × 109/L, platelet count ≥75 × 109/L, hemoglobin ≥ 90g/L, ALB≥30g/L, TBIL ≤30 umol/L, AST ≤5×ULN, ALT ≤5×ULN, ALP ≤5×ULN, Cr ≤1.5×ULN, TSH≤1×ULN and TSH≥LLN, INR≤2.3, prolonged PT≤6s without anticoagulant therapy, urine protein <2+ or urine protein ≥2+ but 24h urine protein quantitative <1.0 g)
10. patients with HBsAg (+) received anti-viral therapy, and patients with HCV-RNA (+) must received anti-viral therapy according to the guidelines and the liver function increases within CTCAE grade 1 during the study
11. Female with fertility must agree to use reliable methods of contraception from the signing of the informed consent until at least 120 days after the last administration of the study drug. And the serum HCG test must be negative within 7 days before the start of the study treatment; and it must be a non-lactating period.
12. For male patients whose partner is a fertile woman, they must agree to use reliable methods of contraception from the signing of the informed consent until at least 120 days after the last administration of the study drug. During the same period of time, male patients must also agree not to donate sperm.

Exclusion Criteria:

1. intrahepatic cholangiocarcinoma, sarcomatoid HCC, mixed cell carcinoma and fibrolamellar cell carcinoma diagnosised by pathology
2. patients with other malignant tumors except HCC within 5 years or at the same time, except for cured localized tumors, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, prostate carcinoma in situ, cervical carcinoma in situ, breast carcinoma in situ, etc.
3. patients who are planning to undergo or have previously received organ or allogeneic bone marrow transplantation
4. history of hepatic encephalopathy
5. moderate and severe ascites with clinical symptoms and uncontrolled pleural effusion and pericardial effusion
6. a history of gastrointestinal bleeding or a clear tendency to gastrointestinal bleeding within 6 months before the start of the study treatment
7. a history of abdominal fistula, gastrointestinal perforation or abdominal abscess occurred within 6 months before the start of study treatment
8. a known hereditary or acquired bleeding (such as coagulopathy) or thrombotic tendency
9. currently using or recently used (within 10 days before the start of the study treatment) anticoagulant drugs
10. thrombosis or embolism occurred within 6 months before the start of study treatment, such as cerebrovascular accident, pulmonary embolism
11. with clinical symptoms or diseases of the heart that are not well controlled
12. suffered from blood pressure that could not be well controlled by antihypertensive medication or a history of hypertensive crisis or hypertensive encephalopathy
13. severe cardiovascular disease occurred within 6 months before the start of study treatment
14. severe, unhealed or dehisced wounds and active ulcers or untreated fractures
15. received major surgery (except for diagnosis) within 4 weeks before the start of the study treatment or is expected to undergo major surgery during the study period
16. unable to swallow pills, malabsorption syndrome, or any condition that affects gastrointestinal absorption
17. a history intestinal obstruction, and/or clinical signs or symptoms of gastrointestinal obstruction that were not relieved after the medical treatment within 6 months before start of the study treatment
18. evidence of intra-abdominal gas that cannot be explained by puncture or recent surgery
19. a history of or current central nervous system metastases
20. a history of or current pulmonary fibrosis, organizing pneumonia and other active pneumonia, or severely impaired lung function, which may interfere with the detection and treatment of suspected drug-related lung toxicity
21. any active autoimmune disease or a history of autoimmune disease which are expected recurrence (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, etc.), except for immune diseases that do not require medical treatment, such as vitiligo, psoriasis, asthma, and well-controlled type I diabetes, etc.
22. patients undergoing immunosuppressive agents or systemic hormone therapy to achieve immunosuppressive purposes, and continues to use it within 2 weeks before signing the informed consent
23. received treatment with a live attenuated vaccine within 28 days before the start of the study treatment, or expected to be vaccinated during camrelizumabtreatment or within 60 days after the last dose of camrelizumab
24. active tuberculosis
25. congenital or acquired immune deficiencies (such as HIV-infected)
26. combined hepatitis B and hepatitis C co-infection
27. patients who are known to be allergic to study drugs or excipients have a history of allergies
28. palliative radiotherapy for non-target lesions for symptom control within 2 weeks before the start of study treatment, or adverse events caused by radiotherapy did not recover to ≤ CTCAE grade 1 (except for alopecia)
29. perform locoreginal treatments of the liver within 28 days before start of the study treatment (such as radiofrequency ablation, percutaneous ethanol or acetic acid injection, cryoablation, high-intensity focused ultrasound, transarterial chemoembolization, transarterial embolization, etc.), or adverse reactions caused by previous locoreginal treatments have not recovered to ≤ CTCAE level 1 (except for alopecia etc.)
30. according to the judgment of the investigator, the patients with factors that may affect the results of the study or cause the study to be terminated midway, such as alcoholism, drug abuse, other serious diseases (including mental illness) need to be treated together, severe laboratory abnormalities, accompanied by family or social factors, which will affect the safety of patients
31. patients who is pregnant or breastfeeding
32. other factors that the investigatior considers inappropriate to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 months
  the The date of randomization to death from any cause

SECONDARY OUTCOMES:
Progression-free survival | 2 months
  The date from randomization until progression according to RECIST 1.1 or death. from any cause
Time to progression | 2 months
  The time from randomization until first evidence of disease progression.
Time to response | 2 months
  The time from initiating treatment to achieve complete or partial response according to RECIST 1.1
Duration of response | 2 months
  The time from randomization to disease progression or death in patients who achieve complete or partial response according to RECIST 1.1
Objective response rate | 2 months
  The proportion of patients with the best response of complete response or partial response according to RECIST 1.1
Disease control rate | 2 months
  The proportion of patients with the best response of complete response, partial response and stable disease according to RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China